CLINICAL TRIAL: NCT01143376
Title: High-intensity Intermittent Training to Maximize Metabolic and Cardiovascular Protection in Obese Individuals
Brief Title: High-intensity Intermittent Training for Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Midt-Norge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/447
Record Dates: First submitted 2010-06-02; First posted 2010-06-14 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Obesity
Keywords: Obesity; exercise; body composition; insulin sensitivity; appetite; food intake
MeSH Terms: conditions — Obesity; Motor Activity; Insulin Resistance | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate intensity exercise (Active Comparator): Moderate intensity exercise
  Interventions: Behavioral: Moderate intensity exercise
- High Intensity training (Experimental): High Intensity intermittent training
  Interventions: Behavioral: High intensity training
- Short springs (Experimental): short springs training
  Interventions: Behavioral: short springs

INTERVENTIONS:
Behavioral: High intensity training — high-intensity intermittent sprinting (HIIS) (8 sec sprint:12 sec rest) for 12 weeks, 4 times a week
  Arms: High Intensity training
Behavioral: short springs — short duration sprints (SDS)(8 sec sprint:12 sec rest) for 12 weeks, 4 times a week
  Arms: Short springs
Behavioral: Moderate intensity exercise
  Arms: Moderate intensity exercise

SUMMARY:
The most appropriate and effective exercise interventions for weight loss remain a matter of continued discussion and there is a need to identify sustainable exercise programs which successfully promote weight loss and benefit health.

The primary objective of this study is to determine if high-intensity intermittent sprinting (HIIS) produces better results in terms of reducing metabolic and cardiovascular risk factors, with special emphasis to fat mass loss and insulin sensitivity in "healthy" obese volunteers compared with an iso-caloric program of moderate-intensity continuous cycling (MICC) (control condition following the international recommendations). We will also assess the impact of short duration sprints (SDS) in the above factors and to understand the potential mechanisms behind different outcomes among training programs.

The overall hypothesis is that HIIS will lead to a greater reduction in metabolic and cardiovascular risk factors compared with MICC in healthy obese volunteers and that SDS will produce similar improvements in cardiovascular risk factors as the longer duration HIIS

DETAILED DESCRIPTION:
Participants will be randomized to one of three groups: HIIS (8s sprint:12s rest) or MICC (control group) iso-caloric protocols (for the duration needed to induce a 250 kcal energy deficit) or SDS (8s sprint:12s rest) for 10 minutes for 12 weeks. The intervention groups will be matched for age, BMI and male/females ratio and participants will be asked not to change their normal diet throughout the study.

Before and after the exercise intervention (12 weeks), participants will perform the following assessments:

1. Three-day food diaries
2. Anthropometric measurements (weight, height, waist and hips) using standard procedures;
3. Body composition using dual energy x-ray absorptiometry (DEXA)
4. RMR and resting respiratory exchange ratio (RER) using indirect calorimetry;
5. Endothelial function assessed by flow-mediated dilation (FMD) of the brachial artery using vascular ultrasound according to current guidelines;
6. Maximal oxygen uptake (VO2max) and fat oxidation, cardiac output and left ventricular function during exercise using a cycle ergometer;
7. Muscle and fat biopsies
8. Fasting and postprandial release of appetite related hormones (and subjective feelings of hunger/fullness using visual analogue scales - VAS).

ELIGIBILITY:
Inclusion Criteria:

* weight stable on the last three months,
* not currently dieting to lose weight
* inactive lifestyle.

Exclusion Criteria:

* History of endocrine/cardiovascular/pulmonary/kidney disease,
* anaemia,
* gout,
* depression or other psychological disorders,
* eating disorders,
* drug or alcohol abuse within the last two years
* current medication known to affect appetite or induce weight loss.
* planned surgery during the study period
* participation in another research study
* restraint score derived from the TFEQ>12
* post-menopausal women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Changes in body composition | Baseline and after 12 weeks of training
  Body composition assessed by DEXA

SECONDARY OUTCOMES:
Changes in insulin sensitivity | Baseline and after 12 weeks of training
  Insulin will be measured in fasting and for 3h after a test meal

CONTACTS AND LOCATIONS:
Overall Officials: Catia Martins, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Martins C, Kazakova I, Ludviksen M, Mehus I, Wisloff U, Kulseng B, Morgan L, King N. High-Intensity Interval Training and Isocaloric Moderate-Intensity Continuous Training Result in Similar Improvements in Body Composition and Fitness in Obese Individuals. Int J Sport Nutr Exerc Metab. 2016 Jun;26(3):197-204. doi: 10.1123/ijsnem.2015-0078. Epub 2015 Oct 19. PMID 26479856
- [Result] Martins C, Aschehoug I, Ludviksen M, Holst J, Finlayson G, Wisloff U, Morgan L, King N, Kulseng B. High-Intensity Interval Training, Appetite, and Reward Value of Food in the Obese. Med Sci Sports Exerc. 2017 Sep;49(9):1851-1858. doi: 10.1249/MSS.0000000000001296. PMID 28398946